CLINICAL TRIAL: NCT06241859
Title: The Influence of Sedation Depth Monitoring for Cognitive Functions and Early Rehabilitation After the Elective Total Knee Joints Replacement Surgery in Elderly Patients: Prospective, Randomized, Double-blind Study
Brief Title: The Impact of Sedation Depth Monitoring for Cognitive Functions and Early Rehabilitation After Major Joints Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Inna Jaremko, MD, Principal investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BE-2-53
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-01

CONDITIONS: Total Knee Replacement Surgery
Keywords: Sedation depth; Cognitive functions; Quality of rehabilitation; Functional recovery; Elective surgery; Total knee arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light sedation according to BIS (Active Comparator): Sedation depth will be monitored according to BIS.
  Interventions: Device: Dräger Infinity Delta series monitor (Dräger, Germany) with Covidien BIS LoC 2 channel module and BIS Quatro (4 electrodes) sensor (Covidien, Ireland)
- Sedation according to clinical signs (Sham Comparator): Sedation depth will be monitored according to clinical signs using RASS scale, which aim is -3.
  Interventions: Device: Dräger Infinity Delta series monitor (Dräger, Germany) with Covidien BIS LoC 2 channel module and BIS Quatro (4 electrodes) sensor (Covidien, Ireland)

INTERVENTIONS:
Device: Dräger Infinity Delta series monitor (Dräger, Germany) with Covidien BIS LoC 2 channel module and BIS Quatro (4 electrodes) sensor (Covidien, Ireland) — Dräger Infinity Delta series monitor (Dräger, Germany) with Covidien BIS LoC 2 channel module and BIS Quatro (4 electrodes) sensor (Covidien, Ireland) will be used to maintain a sedation depth between 80-90 value, which corresponds to light sedation definition.
  Arms: Light sedation according to BIS
Device: Dräger Infinity Delta series monitor (Dräger, Germany) with Covidien BIS LoC 2 channel module and BIS Quatro (4 electrodes) sensor (Covidien, Ireland) — Dräger Infinity Delta series monitor (Dräger, Germany) with Covidien BIS LoC 2 channel module and BIS Quatro (4 electrodes) sensor (Covidien, Ireland) will be used to monitor sedation depth.
  Arms: Sedation according to clinical signs

SUMMARY:
Spinal anesthesia is applied for patients undergoing total elective knee replacement surgery. It reduces rates of postoperative complications, improves postoperative pain management, rehabilitation is started earlier and patients more quickly return to the rhythm of ordinary life. According to the literature data, perioperative stress impacts part of cardiovascular complications and exacerbates postoperative pain. It is important that patients during the surgery under spinal anesthesia prefer to sleep. Thus, in order to reduce perioperative stress, patients during surgery are sedated. It is one of the most effective methods.

On the other hand, deep sedation during surgery versus light sedation, is related to more frequent postoperative cognitive impairment and delirium. It leads to worse later surgery results and worse postoperative quality of life, increased risk of falling, prolonged duration of hospitalization, increased expenses.

DETAILED DESCRIPTION:
The aim: To determine value of sedation depth monitoring in order to save patients cognitive functions, to reduce incidence of postoperative delirium and to improve quality of early rehabilitation after the elective total elective knee replacement surgery.

Primary hypothesis: targeted sedation depth monitoring, in order to support light sedation level during the elective knee arthroplasty, helps to save cognitive function and reduce incident of postoperative delirium.

Secondary hypothesis: targeted sedation depth monitoring, in order to support light sedation level, provide better ability to early rehabilitation and patients more quickly return to the rhythm of ordinary life after elective total knee arthroplasty.

Objectives:

1. To evaluate moderate and deep sedation rates in a group of patients sedated according to clinical signs only.
2. To compare changes in cognitive functions and incidence of delirium after the surgery between a group of patients with light sedation according to bispectral index (BIS) and a group of patients sedated according to clinical signs.
3. To assess the impact of sedation depth monitoring for ability and quality of early rehabilitation after elective total knee replacement surgery.

Methods:

The prospective, randomized, double-blinded study includes American Society of Anesthesiologists (ASA) physical status I-II patients in preoperative assessment, aged >65 years, admitted for the elective total knee arthroplasty under spinal anesthesia with sedation. Preoperatively patients will be blindly randomized into one of two groups. Experimental group: light sedation according to BIS and control group: sedation according to clinical signs. Group assignment will be concealed by opaque envelopes that will be opened only after enrolment. The investigator, who does not interview patients, will document which group the participant belongs to and will provide an unique number. The same investigator will collect data in an operating room. But the participant and outcomes assessor will be blinded to group assignment.

During the perioperative period all patients from both groups will receive a standardized anesthetic and analgesic. Premedication of midazolam 2.5 mg will be given to all patients and a slow fluid infusion of crystalloids will be started once as an intravenous cannula will be placed. Spinal anesthesia after identification of the subarachnoid space will be performed with 15 mg of levobupivacaine. After that, for post operative analgesia femoral triangle and adductor canal blocks will be performed under the ultrasound guidance. Patients will be sedated with intravenously administered propofol according to BIS, in order to support light sedation level (BIS value 80-90), or according to clinical sign (depending on the group of patients) during the surgery. During the surgery BIS and standard monitoring will be performed in both groups. After the surgery patients will be transferred to the post-anesthesia care unit (PACU). During the postoperative period NSAIDs and acetaminophen will be available in both groups.

Patients cognitive function will be evaluated before the surgery and at 2, 30, 90 postoperative days using Addenbrooke's Cognitive Examination test - revised (ACE-R). This is 100-scores test that allows to assess the main six cognitive function domains and weighted as follows: orientation (10), attention (8), memory (26), verbal fluency (14), language (26) and visuospatial ability (16).

The ability and quality of rehabilitation will be assessed before the surgery and at 2, 30, 90 days after the surgery using Quality of Life Questionnaire (SF-36v2 Health Survey). This test allows to assess the main eight quality of life domains: vitality, physical functioning, bodily pain, general health perceptions, role limitations due to physical and emotional health, social rule functioning, mental health.

Patients emotional state will be evaluated using the Geriatric Depression Scale before the surgery and at 2, 30, 90 postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective total knee replacement surgery under spinal anesthesia with sedation;
* Age 66 - 90 years;
* Patients conformed to American Society of Anesthesiologists (ASA) physical status I-II in preoperative assessment;
* Ability to follow study protocol;
* Signed agreement to participate in the study.

Exclusion Criteria:

* Refused elective total knee arthroplasty under spinal anesthesia with sedation;
* Younger than 66 years;
* Patients conformed to American Society of Anesthesiologists (ASA) physical status III-IV in preoperative assessment;
* Patients with mental and central nervous system disorders, which hinder the perception and correct assessment of their condition;
* Hearing, visual, speech disorders and inability to read, write;
* Inability to understand and read in Lithuanian language;
* Refusal to participate in the study.

Ages: 66 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive function using Addenbrooke's Cognitive Examination test | Before the surgery and first 3 months after elective total knee arthroplasty

SECONDARY OUTCOMES:
Quality of functional recovery using the Quality of Life Questionnaire (SF-36v2 Health Survey) | Before the surgery and first 3 months after elective total knee arthroplasty
Rates of moderate and deep sedation according to the BIS in non-interventional group | During the surgery
Changes in emotional state according to geriatric depression scale | Before the surgery and first 3 months after elective total knee arthroplasty

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences Kaunas Clinics, Department of Anesthesiology, Kaunas, Lithuania